CLINICAL TRIAL: NCT00804622
Title: A Randomized, Open-label, Controlled, Exploratory Trial to Characterize the Results of Daily Oral Administration of Telbivudine 600 mg and Tenofovir Disproxil Fumarate 300 mg in Combination or Telbivudine 600 mg or Tenofovir Disproxil Fumarate 300 mg Monotherapy Given Over 12 Weeks on the Kinetics of Hepatitis B Virus DNA in Adults With HBeAg Positive Compensated CHB
Brief Title: Effects of Telbivudine and Tenofovir Disproxil Fumarate on the Kinetics of Hepatitis B Virus DNA in Chronic Hepatitis B (CHB)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Prof. George Lau, Department of Medicine, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLDT600AHK01
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Chronic Hepatitis B
Keywords: HBeAg positive compensated chronic hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Telbivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): tenofovir disproxil fumarate 300 mg monotherapy
  Interventions: Drug: tenofovir disproxil fumarate
- 2 (Active Comparator): telbivudine 600 mg monotherapy
  Interventions: Drug: telbivudine
- 3 (Active Comparator): telbivudine 600 mg and tenofovir disproxil fumarate 300 mg
  Interventions: Drug: telbivudine plus tenofovir disproxil fumarate

INTERVENTIONS:
Drug: telbivudine — daily oral administration,600mg,over 12 weeks
  Arms: 2
Drug: tenofovir disproxil fumarate — daily oral administration,300mg,over 12 weeks
  Arms: 1
Drug: telbivudine plus tenofovir disproxil fumarate — daily oral administration of telbivudine 600 mg and tenofovir disproxil fumarate 300 mg in combination given over 12 weeks
  Arms: 3

SUMMARY:
The purpose of this study is to compare the safety, tolerability and effectiveness of 12 weeks of treatment with telbivudine 600 mg daily plus tenofovir DF 300 mg once daily (QD) taken together versus tenofovir DF 300 mg once daily (QD) or versus telbivudine 600 mg monotherapy daily (QD). This is an open-labeled, active controlled, viral kinetics study which means the subjects and study doctor will know what study drug subjects have been assigned. This study is open to male and female subjects, <40 years of age, who have been infected with HBV for at least 6 months and have not received oral treatment for HBV.

DETAILED DESCRIPTION:
The primary goal of therapy for chronic hepatitis B (CHB) is suppression of viral replication. Long-term suppression of serum HBV DNA is likely to reduce progression to cirrhosis and hepatic decompensation and decrease the risk of hepatocellular carcinoma. Conventional treatment of chronic hepatitis B is limited by low rates of sustained hepatitis B virus DNA suppression and hepatitis B e antigen (HBeAg) seroconversion, increasing rates of drug resistance to the oral agents, and poor tolerability of interferon.

Currently, several nucleoside/nucleotide analogues are available for treatment of CHB. Typically, treatment is continued indefinitely since discontinuation is usually associated with relapse . However, the safety implications related to long term treatment are still unknown.

Previously published studies using combinations (peginterferon alpha-2a + lamivudine) (Marcellin 2004; Lau 2005; Janssen 2005) have shown combinations to be more potent in HBeAg loss at the end of dosing, than either agent used as monotherapy; off-treatment differences, however, did not persist. There are no treatment paradigms as yet of combination therapy with two nucleoside analogues for use in treatment-naive patients.

In summary, there is an unmet need for improved anti-HBV therapy and there are still several controversies such as treatment options, potential role of combination therapy versus monotherapy and optimal duration of therapy, among others. Clinical trials are underway to answer some of these questions. This study aims to assess whether or not combination therapy with telbuvudine and tenofovir DF has superior antiviral efficacy when compared to tenofovir DF or telbuvidine monotherapy. The study will also determine the safety of the combination of telbivudine and tenofovir disoproxil fumarate in patients with chronic hepatitis B. Patients in the immunotolerant phase of CHB will be include in the study. This phase is characterized for high viremia and normal transaminases. Since these patients are not considered as candidates for CHB therapy according to international guidelines (Lok et al 2007), treatment discontinuation after 12 weeks does not raise any unethical implications.

REFERENCES:

1. Janssen HL, van Zonneveld M, Senturk H, Zeuzem S, Akarca US, Cakaloglu Y, Simon C, So TM, Gerken G, de Man RA, Niesters HG, Zondervan P, Hansen B, Schalm SW; HBV 99-01 Study Group; Rotterdam Foundation for Liver Research. Pegylated interferon alfa-2b alone or in combination with lamivudine for HBeAg-positive chronic hepatitis B: a randomised trial. Lancet. 2005 Jan 8-14;365(9454):123-9.
2. Lau GK, Piratvisuth T, Luo KX, Marcellin P, Thongsawat S, Cooksley G, Gane E, Fried MW, Chow WC, Paik SW, Chang WY, Berg T, Flisiak R, McCloud P, Pluck N; Peginterferon Alfa-2a HBeAg-Positive Chronic Hepatitis B Study Group. Peginterferon Alfa-2a, lamivudine, and the combination for HBeAg-positive chronic hepatitis B. N Engl J Med. 2005 Jun 30; 352(26):2682-95.
3. Lok AS, McMahon BJ. (2007) Chronic hepatitis. Hepatology 45(2):507-39.
4. Marcellin P, Lau GK, Bonino F, Farci P, Hadziyannis S, Jin R, Lu ZM, Piratvisuth T, Germanidis G, Yurdaydin C, Diago M, Gurel S, Lai MY, Button P, Pluck N; Peginterferon Alfa-2a HBeAg-Negative Chronic Hepatitis B Study Group. Peginterferon alfa-2a alone, lamivudine alone, and the two in combination in patients with HBeAg-negative chronic hepatitis B. N Engl J Med. 2004 Sep 16;351(12):1206-17.

Primary objectives:

The primary objective of this study is to characterize the reduction in HBV DNA level from Baseline to week 12 of telbivudine plus tenofovir DF combination therapy versus telbivudine or tenofovir DF monotherapy.

Secondary objectives:

Secondary objectives of the study include describing the following for telbivudine plus tenofovir DF combination therapy versus telbivudine or tenofovir DF monotherapy:

1. reduction in HBV DNA level from Baseline to Weeks 2, 4, and 8
2. characterization of early viral kinetics through estimation of various parameters such as efficiency of blocking new virus production, and half-lives of free virions and infected heptocytes
3. % patients who are PCR negative at Week 12 (defined as <25 copies/mL)
4. % of patients who achieve HBeAg loss and HBeAg seroconversion at Week 12
5. safety

Exploratory objectives:

1. To explore HBeAg and HBsAg levels over the treatment period as an additional potential predictor of efficacy.
2. To explore additional potential early serological and immunological markers for prediction of efficacy or safety.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria at screening to be eligible for participation in this study.

1. Chronic HBV infection, defined as positive serum HBsAg for at least 6 months, or HBsAg positive > 3 months and negative for IgM anti-HBc and positive for IgG anti-HBc
2. Age < 40 years old
3. HBeAg positive
4. HBV DNA ≥ 10^7 copies/mL by Abbott real-time PCR
5. ALT ≤ 1 ULN
6. Willing and able to provide written informed consent
7. Negative serum β-HCG (for females of childbearing potential only)
8. Calculated creatinine clearance ≥ 70 mL/min by the following formula: (140 - age in years) x (body weight [kg]) / (72) x (serum creatinine [mg/dl]) [Note: multiply estimated rate by 0.85 for women]
9. Hemoglobin ≥ 10 g/dL
10. Neutrophils ≥ 1,500 /mm^3
11. No prior oral HBV therapy (e.g., nucleotide and/or nucleoside therapy or other investigational agents for HBV infection)
12. Is willing and able to comply with the study drug regimen and all other study procedures and requirements
13. Is willing and able to provide written informed consent before any study assessment is perform.

Exclusion Criteria:

Patients will be excluded from the study for any of the criteria:

1. Decompensated liver disease defined as direct (conjugated) bilirubin > 1.2 × ULN, PT > 1.2 × ULN, platelets < 150,000/mm3, serum albumin < 3.5 g/dL, or prior history of clinical hepatic decompensation (e.g. ascites, jaundice, encephalopathy, variceal hemorrhage).
2. Received interferon (pegylated or not) therapy within 6 months of the screening visit
3. α-fetoprotein > 50 ng/mL
4. Evidence of hepatocellular carcinoma (HCC)
5. Co-infection with HCV (by serology), HIV, or HDV.
6. Significant renal, cardiovascular, pulmonary, or neurological disease.
7. Received solid organ or bone marrow transplantation.
8. Is currently receiving therapy with immunomodulators (e.g., corticosteroids, etc.), investigational agents, nephrotoxic agents, or agents susceptible of modifying renal excretion.
9. Has proximal tubulopathy.
10. Use of other investigational drugs at the time of enrollment, or within 30 days
11. History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes
12. Is pregnant or breastfeeding. Women of childbearing potential must have a negative serum β - HCG during Screening.
13. Is a women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner and women whose partners have been sterilized by vasectomy or other means, UNLESS they meet the following definition of post-menopausal: 12 months of natural (spontaneous) amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels >40 mIU/m or 6 weeks post surgical bilateral oophorectomy with or without hysterectomy OR are using one or more of the following acceptable methods of contraception: surgical sterilization (e.g., bilateral tubal ligation, vasectomy), hormonal contraception (implantable, patch, oral), and double-barrier methods (any double combination of: IUD, male or female condom with spermicidal gel, diaphragm, sponge, cervical cap).
14. Patient has any other concurrent medical or social condition likely to preclude compliance with the schedule of evaluations in the protocol, or likely to confound the efficacy or safety observations of the study.
15. Patient is currently abusing alcohol or illicit drugs, or has a history of alcohol abuse or illicit substance abuse within the preceding two years. Please refer to Appendix 3.
16. Patient has a medical condition that requires prolonged or frequent use of systemic acyclovir or famciclovir. Please refer to Appendix 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-12; Primary Completion 2009-06 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
The primary variable is the reduction of HBV DNA level over 12 weeks of treatment | 12 weeks

SECONDARY OUTCOMES:
Reduction in HBV DNA level | from baseline to Weeks 2, 4 and 8
Characterization of very early viral kinetics through estimation of various parameters | week 12
% patients who are PCR negative | Week 12
% of patients who achieve HBeAg loss and HBeAg seroconversion | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: George Lau, MD, Principal Investigator — Department of Medicine, The University of Hong Kong
Locations (1):
- Department of Medicine, Queen Mary Hospital, Hong Kong, China